CLINICAL TRIAL: NCT03129802
Title: Incidence and Risk Factors of Extubation Failure in Pediatric Resuscitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6310
Record Dates: First submitted 2016-06-17; First posted 2017-04-26 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2016-06

CONDITIONS: Respiratory Insufficiency
Keywords: extubation; pediatric resuscitation; reintubation; failures of extubation.; Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The failure of extubation in pediatric resuscitation is most often described as the need for reintubation within 48 hours after extubation. The failure rate of extubation in pediatric intensive care varies in the literature there is 4 to 22% failure. These failures result in increased mortality, morbidity with a use of larger tracheostomy, a prolonged residence time. Some risk factors are well defined in the literature as the duration of intubation, ENT and neurological history, the persistence of a respiratory disease, a high level of sedation. Other factors are more controversial as age, ventilatory parameters just before extubation before extubation blood gases, the interest of a leak test.

Also pediatric populations are extremely heterogeneous, so the investigators would like to highlight to extubation failure risk factors in Hautepierre pediatric ICU to better support these high-risk children.

ELIGIBILITY:
Inclusion Criteria:

* Children hospitalized in pediatric intensive care, under 18 years, intubated, ventilated for more than 2 hours and for which planning extubation or intubated children for whom an unplanned extubation just happened.
* Children whose holding parental authority are not opposed to the use of clinical data from their child for research purposes.

Exclusion Criteria:

* Refusal to participate in the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children hospitalized in pediatric intensive care, under 18 years, intubated, ventilated for more than 2 hours and for which planning extubation or intubated children for whom an unplanned extubation just happened.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Failure of extubation | need for a new intubation within the first 48 hours after extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Reanimation Pediatrique Specialisee - S. Continue, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No